CLINICAL TRIAL: NCT00162370
Title: SMART: Stress Echocardiography in Menopausal Women at Risk for Coronary Artery Disease Trial
Brief Title: A Study of Stress Echocardiography in Post-Menopausal Women at Risk for Coronary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMP 115-407
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease; Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Definity (Experimental): All patients will undergo a gray scale baseline unenhanced imaging session (apical 2- or 4 chamber view), as well as a DEFINITY (Perflutren Lipid Microsphere Injectable Suspension)-enhanced rest and a DEFINITY enhanced exercise or dobutamine stress echocardiography imaging session. The unenhanced and DEFINITY-enhanced rest and stress echocardiography imaging sessions will be performed on the same day. For the DEFINITY-enhanced imaging sessions all patients will receive diluted DEFINITY intravenously (IV). Diluted DEFINITY will be prepared by mixing 1 mL of activated DEFINITY® with 9 mL of normal saline in a 10 mL syringe.
  Interventions: Drug: Perflutren Lipid Microsphere Injectable Suspension

INTERVENTIONS:
Drug: Perflutren Lipid Microsphere Injectable Suspension — Activated DEFINITY 10ug/kg by bolus injection
  Other Names: DEFINITY

SUMMARY:
The study is designed to see if stress echocardiography can be used as a screening exam in peri-, or post-menopausal women with a risk of developing of coronary artery disease and experiencing future cardiac events.

DETAILED DESCRIPTION:
The clinical trial is designed to determine the prognostic value of stress echocardiography as a screening examination in peri-, or post-menopausal female patients with an intermediate likelihood of coronary artery disease (CAD) based on risk factors to identify patients at higher risk of experiencing future cardiac events.Female patients who are able to adequately exercise will undergo a symptom-limited exercise echocardiogram. Patients who are unable to adequately exercise or are predicted to be unable to exercise adequately (because of orthopedic/neurologic limitations, lung disease or debility), will perform dobutamine stress echocardiography. All patients will receive DEFINITY at rest and stress to enhance wall motion assessment.

ELIGIBILITY:
Inclusion Criteria:

* Peri or Post menopausal women either:

  * without symptoms but with risk factors for heart disease OR
  * experiencing atypical chest pain, OR
  * experiencing exertional dyspnea AND 2 or more risk factors for CAD
* Must be able to perform an exercise stress test

Peri-or post-menopausal (including surgical menopause) based on history.

* Post-menopausal is defined as females age 40-65 who self-report the absence of menstrual periods for at least 12 months.
* Peri-menopausal is defined as females age 40-65 who self-report the absence or irregularity of menstrual periods for 6-12 months.
* Surgical menopause is defined as females who have had a bilateral salpingo-oophorectomy with or without hysterectomy.

Exclusion Criteria:

* Previous confirmed heart disease

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-04; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Mulvagh, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Local Institution, Scottsdale, Arizona
  - Local Institution, Jacksonville, Florida
  - Local Institution, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelmoneim SS, Ball CA, Mantovani F, Hagen ME, Eifert-Rain S, Wilansky S, Castello R, Pellikka PA, Best PJM, Mulvagh SL. Prognostic Utility of Stress Testing and Cardiac Biomarkers in Menopausal Women at Low to Intermediate Risk for Coronary ARTery Disease (SMART Study): 5-Year Outcome. J Womens Health (Larchmt). 2018 May;27(5):542-551. doi: 10.1089/jwh.2017.6506. Epub 2018 Apr 19. PMID 29672210
- [Derived] Mantovani F, Abdelmoneim SS, Zysek V, Eifert-Rain S, Mulvagh SL. Effect of stress echocardiography testing on changes in cardiovascular risk behaviors in postmenopausal women: a prospective survey study. J Womens Health (Larchmt). 2014 Jul;23(7):581-7. doi: 10.1089/jwh.2013.4604. Epub 2014 Jun 16. PMID 24932797

RESULTS

PARTICIPANT FLOW:
Groups:
- Definity: Open-lable, non-randomized, Phase IV trial with Definity to determine the prognostic value of stress echocardiogrophy as a screening exam in peri-, post-menopausal females with an intermediate likelihood of coronary artery disease to identify patients at higher risk of experiencing future cardiac events.
  Perflutren Lipid Microsphere Injectable Suspension: Activated DEFINITY 10ug/kg by bolus injection
Period: Completed Echocardiography Imaging
Arm/Group | Definity
Started | 366 (Received at least one dose of Definity)
Completed | 366 (number of subjects who under went Definity-enhanced rest and stress echocardiogram)
Not Completed | 0
Period: Efficacy Population
Arm/Group | Definity
Started | 366
Completed | 315 (Efficacy population, completed rest/stress echo with Definity & completed 2 and/or 5 year follow up)
Not Completed | 51
Not completed — Lost to Follow-up | 51

BASELINE CHARACTERISTICS:
Population: Peri- or post-menopausal female subjects between 40 and 65 years of age with an intermediate likelihood of CAD who are scheduled to undergo stress echocardiography
Groups:
- Definity: Open-label, non-randomized, Phase IV trial with Definity to determine the prognostic value of stress echocardiogrophy as a screening exam in peri-, post-menopausal females with an intermediate likelihood of coronary artery disease to identify patients at higher risk of experiencing future cardiac events.
  Perflutren Lipid Microsphere Injectable Suspension: Activated DEFINITY 10ug/kg by bolus injection
Arm/Group | Definity
Number analyzed (Participants) | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 394
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: Years] | 54.4 [40 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 400
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 386
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 400

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormal Contrast Stress Echocardiography and With Future Major Adverse Cardiac Events (MACE) at 2 and 5 Years Follow-Up
Description: Peri- or post-menopausal female participants with an intermediate pre-test likelihood of coronary artery disease (CAD) received a Definity contrast-enhanced stress echocardiography study at baseline using either treadmill exercise or dobutamine stresss. Images were evaluated for wall motion abnormalities. The results were compared to patient history on 2-year and 5-year follow up to identify the potential of stress echocardiography for predicting those at higher risk of experiencing future cardiac events.
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 2 year and 5 year follow up
Population: Subject has received a physical exam, completed patient history profile, undergone the protocol-specific unenhanced and DEFINITY enhanced rest and stress echocardiography, had the necessary blood work for the study and participated in 2 year or 5 year follow up
Measure: Count of Participants; unit: Participants
Groups:
- Definity: Open-label, non-randomized, Phase IV trial with Definity to determine the prognostic value of stress echocardiogrophy as a screening exam in peri- and post-menopausal females with an intermediate likelihood of coronary artery disease to identify patients at higher risk of experiencing future cardiac events.
  Perflutren Lipid Microsphere Injectable Suspension: Activated DEFINITY 10ug/kg by bolus injection
Arm/Group | Definity
Number analyzed (Participants) | 363
Participants
  Abnormal contrast stress echo and any major cardiac event at 2 year follow up: number analyzed (Participants) | 43
  Abnormal contrast stress echo and any major cardiac event at 2 year follow up | 2
  Normal contrast stress echo and any major cardiac event at 2 year follow up: number analyzed (Participants) | 320
  Normal contrast stress echo and any major cardiac event at 2 year follow up | 1
  Abnormal contrast stress echo and any major cardiac event at 5 year follow up: number analyzed (Participants) | 43
  Abnormal contrast stress echo and any major cardiac event at 5 year follow up | 1
  Normal contrast stress echo and any major cardiac event at 5 year follow up: number analyzed (Participants) | 320
  Normal contrast stress echo and any major cardiac event at 5 year follow up | 5
Statistical Analysis 1: Comparison: Definity; The null hypothesis evaluated is that the scores are not associated with outcome. Of the two measures, wall motion index is considered to be the primary endpoint measure. The cardiac event rate will be summarized by categorical levels of wall motion index score and the difference in wall motion index score; Test type: Superiority or Other; p = 0.014, Regression, Cox

2. Secondary Outcome: Number of Participants With Abnormal ECG and With Major Adverse Cardiac Events (MACE) at 2 Year Follow-Up
Description: Prognostic value of stress ECG testing for identifying female patients at increased risk of major adverse cardiac events (MACE) at 2-year follow-up
  Peri- or post-meopausal female subjects with an intermediate pre-test likelihood of coronary artery disease (CAD) received resting ECG at baseline. ECG was evaluated as normal or abnormal. The results were compared to patient history on 2-year follow up to identify the potential for ECG to predict those at higher risk of experiencing future cardiac events.
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 2-year follow-up
Population: Subject has received a physical exam, completed patient history profile, undergone the protocol-specific unenhanced and DEFINITY enhanced rest and stress echocardiography, had the necessary blood work for the study and participated in 2 year follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Definity
Number analyzed (Participants) | 18
Participants
  Number of subjects with abnormal stress ECG at baseline who had MACE at 2 years | 3
  Number of subjects with abnormal stress ECG at baseline who did not have MACE at 2 years | 15
Statistical Analysis 1: Comparison: Definity; Test type: Superiority or Other; p < 0.0001, Regression, Cox

3. Secondary Outcome: Change in Brain Natriuretic Peptide (BNP) in Subjects With and Without Major Adverse Cardiac Events at 2-year Follow-up.
Description: The value of exercise-induced changes in blood concentration of cardiac peptide, brain natriuretic peptide (BNP in pg/mL in blood), was assessed in identifying patients with cardiac events at 2-year follow-up. The change in mean BNP blood concentration from rest to stress at baseline is summarized using number of subjects with and without MACE at 2-year follow-up
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 2 year follow up
Population: Participants with valid BNP measurements at both rest and stress and who participated in 2-year follow up
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Definity
Number analyzed (Participants) | 236
pg/mL
  Change of BNP from rest to stress in subjects without major cardiac events at 2 year followup: number analyzed (Participants) | 233
  Change of BNP from rest to stress in subjects without major cardiac events at 2 year followup | 5.2 [0.61 to 9.79]
  Change of BNP from rest to stress in subjects with major cardiac events at 2 year followup: number analyzed (Participants) | 3
  Change of BNP from rest to stress in subjects with major cardiac events at 2 year followup | 10.7 [-32.5 to 53.9]

4. Secondary Outcome: Change in Atrial Natriuretic Peptide (ANP) in Subjects With and Without Major Adverse Cardiac Events at 2-year Follow-up.
Description: The value of exercise-induced changes in blood concentration of cardiac peptide, atrial natriuretic peptide (ANP in pg/mL in blood), was assessed in identifying patients with cardiac events at 2-year follow-up. The change in mean ANP blood concentration from rest to stress at baseline is summarized using number of subjects with and without major adverse cardiac events (MACE) at 2-year follow-up.
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 2 year follow up
Population: Participants with valid ANP measurements at both rest and stress who participated in 2-year follow up
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Definity
Number analyzed (Participants) | 179
pg/mL
  Change of ANP from rest to stress in subjects without major cardiac events at 2-year follow-up: number analyzed (Participants) | 177
  Change of ANP from rest to stress in subjects without major cardiac events at 2-year follow-up | 5.9 [-98.81 to 110.61]
  Change of ANP from rest to stress in subjects with major cardiac events at 2-year follow-up: number analyzed (Participants) | 2
  Change of ANP from rest to stress in subjects with major cardiac events at 2-year follow-up | 101 [-716.32 to 918.32]

5. Secondary Outcome: Change in Brachial Artery Reactivity Was Assessed in in a Subset of Participants With and Without Major Adverse Cardiac Events at 2-year and 5-year Follow-up.
Description: A subset of the study population of peri- or post-meopausal female participants with an intermediate pre-test likelihood of coronary artery disease (CAD) was assessed for brachial artery reactivity at baseline. Brachial diameter was assessed using ultrasound and a pressure cuff both before and after administration of sublingual nitroglycerin. The results were compared to patient history on 2-year and 5-year follow up to identify the potential for brachial artery reactivity to predict those at higher risk of experiencing future cardiac events.The brachial artery reactivity was summarized using number of subjects with and without MACE on follow-up.
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 2 year and 5 year follow up
Population: Subjects with valid brachial artery diameter asurements at both rest and stress. Note that among the subjects in the trial who had MACE either at 2 year or 5 years, none had been assessed for brachial artery reactivity.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Definity
Number analyzed (Participants) | 11
Percentage
  Mean %change of brachial artery diameter from rest to stress in subjects w/o MACE at 2 year followup: number analyzed (Participants) | 5
  Mean %change of brachial artery diameter from rest to stress in subjects w/o MACE at 2 year followup | 7.8 [4.33 to 11.27]
  Mean %change of brachial artery diameter from rest to stress in subjects w/MACE at 2 year followup: number analyzed (Participants) | 0
  Mean %change of brachial artery diameter from rest to stress in subjects w/o MACE at 5 year followup: number analyzed (Participants) | 6
  Mean %change of brachial artery diameter from rest to stress in subjects w/o MACE at 5 year followup | 7.3 [4.32 to 10.28]
  Mean %change of brachial artery diameter from rest to stress in subjects w/MACE at 5 year followup: number analyzed (Participants) | 0

6. Secondary Outcome: Mean Baseline Calcium Score of Participants With and Without Major Cardiac Events at 2-year Follow up.
Description: Coronary artery calcium scoring assesses calcification of the coronary arteries using electron-beam computed tomography (EBCT). It is a sum of lesion scores of area and density above a threshold density. There is no intrinsic upper limit to the calcium score but values above 1000 may not be measurable.
  A subset of peri- or post-meopausal females with an intermediate pre-test likelihood of coronary artery disease (CAD) received resting EBCT at baseline. Images were evaluated for calcium score and results compared to patient history on 2-year follow up, Mean calcium score with confidence interval was summarized for subjects with and without major cardiac events (MACE) at 2-year follow up.
  Calcium score for general population:
  Score Description Relative Risk 0 No evidence of CAD 0 1-112 Average Risk of CAD 1.9 100-400 Moderate risk of CAD 4.3 400-999 High risk of CAD 7.2 1000 Very high risk of CAD 10.8
Time Frame: 2 year follow up
Population: Participants with EBCT-based calcium score assessment at baseline who participated in 2-year follow up
Measure: Mean (95% Confidence Interval); unit: score on a scale (calcium score)
Arm/Group | Definity
Number analyzed (Participants) | 82
score on a scale (calcium score)
  Mean calcium score of subjects without major cardiac events at 2 year follow-up | 45 [16.51 to 73.49]
  Mean calcium score of subjects with major cardiac events at 2 year follow-up: number analyzed (Participants) | 0

7. Secondary Outcome: The Presence of Wall Motion Abnormalities on Definity Stress Echocardiography Assessed for Participants With Both Normal and Abnormal Angiography
Description: In the sub-set of efficacy-evaluable participants who underwent clinically indicated coronary angiography, the accuracy of exercise echocardiography vs. angiography was determined for the detection of CAD. Positive angiography was defined as any stenosis greater than or equal to 50% in any vessel. Wall motion index change indicating abnormal motion was defined as greater than or equal to 13% in 2 or more segments. Angiography was required to have taken place within 60 days following stress echocardiography.
Time Frame: 60 days
Population: Subjects who underwent both rest and stress Definity-enhanced echocardiography and coronary angiography within 60 days
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Undergoing Clinically-indicated Angiography: Subset of the enrolled population who underwent angiography as part of their care.
Arm/Group | Subjects Undergoing Clinically-indicated Angiography
Number analyzed (Participants) | 24
Participants
  Subjects w/negative coronary angiography w/o Definity-enhanced stress echo wall motion abnormality | 7
  Subjects w/negative coronary angiography with Definity-enhanced stress echo wall motion abnormality | 12
  Subjects w/positive coronary angiography w/o Definity-enhanced stress echo wall motion abnormality | 1
  Subjects w/positive coronary angiography and Definity-enhanced stress echo wall motion abnormality | 4

8. Secondary Outcome: Participants With Positive and Negative Angiography Compared With Their ECG Results
Description: In the sub-set of efficacy-evaluable participants who underwent clinically indicated coronary angiography, the accuracy of exercise ECG vs. angiography was determined for the detection of CAD. Positive angiography was defined as any stenosis greater than or equal to 50% in any vessel.
Time Frame: 60 days
Population: Subjects who underwent exercise ECG testing and coronary angiography within 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Undergoing Clinically-indicated Angiography
Number analyzed (Participants) | 24
Participants
  Subjects negative coronary angiography and negative ECG | 15
  Subjects negative coronary angiography and positive ECG | 4
  Subjects w/positive coronary angiography and negative ECG | 3
  Subjects w/positive coronary angiography and positive ECG | 2

9. Secondary Outcome: Number of Participants With Abnormal ECG and With Future Major Adverse Cardiac Events (MACE) at 5 Years Follow-Up
Description: Prognostic value of stress ECG testing for identifying female patients at increased risk of major adverse cardiac events (MACE) at 5-year follow-up
  Peri- or post-meopausal female participants with an intermediate pre-test likelihood of coronary artery disease (CAD) received resting ECG at baseline. ECG was evaluated as normal or abnormal. The results were compared to patient history on 5-year follow up to identify the potential for ECG to predict those at higher risk of experiencing future major adverse cardiac events (MACE) at 5-year follow up.
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 5 year follow up
Population: Subject has received a physical exam, completed patient history profile, undergone the protocol-specific unenhanced and DEFINITY enhanced rest and stress echocardiography, had the necessary blood work for the study and 2 and/or 5 year follow up
Measure: Number; unit: Percent of participants
Arm/Group | Definity
Number analyzed (Participants) | 265
Percent of participants
  Percent of subjects with abnormal stress ECG at baseline who had MACE at 5 years | 16.7
  Percent of subjects with abnormal stress ECG at baseline who did not have MACE at 5 years | 5.0

10. Secondary Outcome: Change in Brain Natriuretic Peptide (BNP) in Participants With and Without Major Adverse Cardiac Events at 5-year Follow-up.
Description: The value of exercise-induced changes in blood concentration of the cardiac peptide, brain natriuretic peptide (BNP in pg/mL in blood), was assessed in identifying patients with cardiac events at 5-year follow-up. The change in mean BNP blood concentration at baseline from rest to stress is summarized using number of participants with and without MACE at 5-year follow up.
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 5 year follow up
Population: Subjects with valid BNP measurements at both rest and stress
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Definity
Number analyzed (Participants) | 234
pg/mL
  Change of BNP from rest to stress in subjects without major cardiac events at 5 year followup: number analyzed (Participants) | 230
  Change of BNP from rest to stress in subjects without major cardiac events at 5 year followup | 4.9 [0.28 to 9.52]
  Change of BNP from rest to stress in subjects with major cardiac events at 5 year followup: number analyzed (Participants) | 4
  Change of BNP from rest to stress in subjects with major cardiac events at 5 year followup | 4.1 [-11.89 to 20.09]

11. Secondary Outcome: Change in Atrial Natriuretic Peptide (ANP) in Participants With and Without Major Adverse Cardiac Events at 5-year Follow-up.
Description: The baseline value of exercise-induced changes in blood concentration of the cardiac peptide, atrial natriuretic peptide (ANP in pg/mL in blood), was assessed in identifying patients with cardiac events at 5-year follow-up. The change in mean ANP blood concentration from rest to stress at baseline was summarized using number of subjects with and without major adverse cardiac events (MACE) at 5-year follow up.
  Major adverse cardiac events (MACE) are defined as
  * Cardiac death
  * Myocardial infarction
  * Cardiac revascularization (PCI or CABG)
  * Hospitalization for chest pain or to rule out myocardial infarction
  * Development of typical angina
  * Development of heart failure
Time Frame: 5 year follow up
Population: Subjects with valid ANP measurements at both rest and stress and follow up at 5 years
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Definity
Number analyzed (Participants) | 178
pg/mL
  Change of ANP from rest to stress in subjects without major cardiac events at 5-year follow-up: number analyzed (Participants) | 174
  Change of ANP from rest to stress in subjects without major cardiac events at 5-year follow-up | -37.4 [-165.64 to 90.84]
  Change of ANP from rest to stress in subjects with major cardiac events at 5-year follow-up: number analyzed (Participants) | 4
  Change of ANP from rest to stress in subjects with major cardiac events at 5-year follow-up | 70.5 [-471.2 to 612.2]

12. Secondary Outcome: Mean Calcium Score of Participants With and Without Major Cardiac Events at 5-year Follow up.
Description: Coronary artery calcium scoring assesses calcification of the coronary arteries using electron-beam computed tomography (EBCT). It is a sum of lesion scores of area and density above a threshold density. There is no intrinsic upper limit to the calcium score but values above 1000 may not be measurable.
  A subset of peri- or post-meopausal females with an intermediate pre-test likelihood of coronary artery disease (CAD) received resting EBCT at baseline. Images were evaluated for calcium score and results compared to patient history on 5-year follow up, Mean calcium score with confidence interval was summarized for subjects with and without major cardiac events (MACE) at 5-year follow up
  Calcium score for general population:
  Score Description Relative Risk 0 No evidence of CAD 0 1-112 Average Risk of CAD 1.9 100-400 Moderate risk of CAD 4.3 400-999 High risk of CAD 7.2 1000 Very high risk of CAD 10.8
Time Frame: 5 year follow up
Population: Participants with EBCT-based calcium score assessment at baseline who participated in 5-year follow up
Measure: Mean (95% Confidence Interval); unit: score on a scale (calcium score)
Arm/Group | Definity
Number analyzed (Participants) | 91
score on a scale (calcium score)
  Mean calcium score of subjects without major cardiac events at 5 year follow-up: number analyzed (Participants) | 90
  Mean calcium score of subjects without major cardiac events at 5 year follow-up | 40.2 [14.52 to 65.88]
  Mean calcium score of subjects with major cardiac events at 5 year follow-up: number analyzed (Participants) | 1
  Mean calcium score of subjects with major cardiac events at 5 year follow-up | 100 [NA to NA] — As there was only one participant in this category, a confidence interval could not be calculated

ADVERSE EVENTS:
Arm/Group | Definity
Serious Adverse Events (participants affected / at risk) | 0/400
Other Adverse Events (participants affected / at risk) | 6/400
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Definity (N=400)
Back Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urticaria NOS (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less